CLINICAL TRIAL: NCT02221778
Title: Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma Patients With Partial Response to Transarterial Chemoembolization
Brief Title: SBRT for Hepatocellular Carcinoma Patients With Partial Response to TACE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre Tsin Chih Chen, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-02/2014
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular; SBRT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBRT (Experimental): SBRT according to the intervention description
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT will be prescribed according to the Radiation Therapy Oncology Group (RTOG) 1112 protocol using Mean Liver Dose (MLD) as parameter. MLD will be calculated using Liver minus Gross Tumor Volume (GTV). Prescription dose will follow the scheme below:
  Prescription dose(Gy) / (MLD) (Gy)
  50 / 13
  45 / 15
  40 / 15
  35 / 15.5
  30 / 16
  27.5 / 17
  If the dose constraints cannot be met, prescription will be according to the level immediately bellow.
  Treatment will be delivered in 5 fractions in consecutive working days

SUMMARY:
This is a pilot study where patients with Hepatocellular Carcinoma (HCC) that have failed Transarterial Chemoembolization (TACE) will be treated with Stereotactic Body Radiation Therapy (SBRT). The focus of the study will be to evaluate safety and efficacy in our population of patients.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosis according to the American Association for the Study of Liver Diseases (AASLD) 2010 criteria
* Tumor Stage
* liver only disease
* tumor thrombus at segment is allowed
* no extra hepatic metastases
* tumor encompassing less than 50% of hepatic volume
* previous treatment with Transarterial Chemo Embolization (TACE) - patient must have performed at least 2 sessions of TACE and have signs of viable tumor in CT or MRI performed 30-40 days after last TACE
* presence of measurable lesion (at least one lesion that can be measured equal or more than 1 cm in CT or MRI).
* Maximum lesion size of 10 cm.
* Liver residual volume equal or more than 700cc or 40% of total liver volume
* Child-Pugh A or absence of hepatic cirrhosis
* absence of encephalopathy or ascitis on clinical exam
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Lab exams:
* hemoglobin > or equal 8 mg/dl
* neutrophils > or equal 1.200/mm³
* platelets > or equal 45.000/mm³
* alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 6 times the upper normal limit
* bilirubin equal or < 2 mg/dl
* international normalized ratio (INR) < 1.7
* serum creatinine equal or < 1.5 times the upper normal limit or creatinine clearance > or equal 60 ml/min
* Albumin >2.8 mg/dl
* not being pregnant - a negative pregnancy test is required (for women). Patients in fertile age should use a contraceptive method during treatment and 4 months after.

Exclusion Criteria:

* Patients with more than 5 discrete lesions in the liver
* Main or common biliary duct invasion
* Patients with main portal vein tumor thrombus or more than 2 portal branch thrombus
* Patients in systemic treatment (sorafenib, chemotherapy). There should be an interval of at least 4 weeks between any medication for treatment of HCC and the current study treatment
* Previous radiation to upper abdomen
* Patients with other malignant neoplasms or previous malignant neoplasms will be accepted in the study if HCC prognosis is worse
* Patients with ischemic myocardial infarction within the last 6 months
* Patients with large esophageal varices with red color sign or bleeding within the last 3 months
* Patients with symptoms of colitis, enteritis, esophagitis, fistula, ileus, necrosis, stenosis or ulcer
* Patients with severe anorexy, constipation, dehydration, diarrhea or vomiting
* Patients unable to understand and sign written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Local Progression Free Survival | 5 years
  Local Progression Free Survival will be measured on triphasic Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) when clinically indicated.
  The exam will be performed every 3 months after the end of treatment. The tumor response will be measured according to the modified RECIST (mRECIST) directed to the HCC study.
  Local Progression Free Survival will be defined as increase of 20% in the sum of all diameters of the treated lesions.
  Time-to-event will be counted from the initiation of SBRT

SECONDARY OUTCOMES:
Distant Progression Free Survival | 5 years
  Distant Progression Free Survival will be measured on triphasic Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) when clinically indicated.
  The exam will be performed every 3 months after the end of treatment. The tumor response will be measured according to the modified RECIST (mRECIST) directed to the HCC study.
  Distant Progression Free Survival will be defined as the appearance of a new hepatic lesion, tumoral thrombus or distant metastases.
  Time-to-event will be counted from the initiation of SBRT
Toxicity | 5 years
  Toxicity will be evaluated according to the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v.4.0). Toxicity will be evaluated weekly during treatment, monthly in the first 3 months after treatment and every 3 months after.
  Acute Toxicity will be defined as toxicity that develops within the first 3 months after initiation treatment.
  Chronic Toxicity will be defined as toxicity that develops after 3 months of initiation of treatment.
Overall Survival | 5 years
  Time-to-event will be counted from the initiation of SBRT

CONTACTS AND LOCATIONS:
Overall Officials: Flair J Carrilho, MD, PhD, Study Chair — University of Sao Paulo; Andre T Chen, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil

REFERENCES:
- [Derived] Chen ATC, Payao F, Chagas AL, De Souza Melo Alencar RS, Tani CM, da Conceicao Vasconcelos KGM, de Souza Rocha M, de Andrade Carvalho H, Hoff PMG, Carrilho FJ. Feasibility of SBRT for hepatocellular carcinoma in Brazil - a prospective pilot study. Rep Pract Oncol Radiother. 2021 Apr 14;26(2):226-236. doi: 10.5603/RPOR.a2021.0035. eCollection 2021. PMID 34211773